CLINICAL TRIAL: NCT02253797
Title: A Phase I Multiple Oral Dose Trial of Tipranavir 500 mg/Ritonavir 200 mg Dosed to Steady State Followed by Single-dose 14C-radiolabeled Tipranavir Co-administered With Tipranavir 500 mg/Ritonavir 200 mg to Characterize the Excretion Balance and Metabolite Profile of 14C-radiolabeled Tipranavir in Healthy Male Subjects
Brief Title: Pharmacokinetics of Tipranavir/Ritonavir and Its Metabolites in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.24
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir

ARMS (1):
- TPV/r followed by 14C-radiolabeled TPV (Experimental): Tipranavir/Ritonavir dosed to steady state followed by single-dose 14C-radiolabeled tipranavir co-administered with Tipranavir/Ritonavir
  Interventions: Drug: 14C-Tipranavir; Drug: Tipranavir; Drug: Ritonavir

INTERVENTIONS:
Drug: 14C-Tipranavir
Drug: Tipranavir
Drug: Ritonavir

SUMMARY:
Study to evaluate the pharmacokinetics of Tipranavir and its metabolites including excretion and mass balance of parent compound and radioactivity at steady-state; to isolate, identify and quantify major metabolites of tipranavir in plasma, urine and feces

ELIGIBILITY:
Inclusion Criteria:

1. Healthy HIV-negative male subjects as determined by results of screening. Healthiness was determined by medical history, laboratory testing and 12-lead ECG
2. Signed written informed consent in accordance with Good Clinical Practice (GCP)
3. Age >18 and <=60 years
4. Subjects within 20% of the normal height: weight range defined by the Metropolitan Life Insurance Company Tables
5. Ability to swallow numerous large capsules
6. Willingness to abstain from smoking, ingesting methylxanthine containing drinks or food (coffee, tea, cola, chocolate, etc.), or ingesting alcohol, St. John's Wort, milk thistle, garlic supplements, Seville oranges, and grapefruit or grapefruit juice for the duration of the study

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate, and ECG) deviating from normal and of clinical relevance
2. History of clinically significant disease including metabolic, endocrinologic, immunological, hepatic, renal, gastrointestinal, respiratory, cardiovascular, psychiatric or neurological
3. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator and/or the sponsor
4. Subjects with a history of drug abuse or alcoholism
5. Chronic or relevant acute (within 2 weeks of screening) infections
6. Subjects who have taken prescription medications, over-the-counter drugs, or herbal preparations within 2 weeks of the start of the trial
7. Participation in another trial with an investigational drug (in the 30 days prior to screening)
8. Blood donation >400 mL (within 1 month prior to treatment administration or during the trial)
9. Any laboratory value that represents a Division of DAIDS (DAIDS) toxicity Grade >1
10. Positive urine drug screen, positive HIV antibody, positive Hepatitis C Ribonucleic acid (RNA), or positive Hepatitis B surface antigen
11. History of any familial bleeding disorder

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-07; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Radioactive levels of 14C-Tipranavir in plasma and blood | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
Radioactive erythrocyte-plasma partition ratio | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
Maximum measured concentration of the analyte in plasma (Cmax) | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
  14C-radiolabeled Tipranavir + Tipranavir
Plasma concentration 12 hours after dosing (Cp12h) | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
  14C-radiolabeled Tipranavir + Tipranavir
Area under plasma concentration time curve (AUC) | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
  14C-radiolabeled Tipranavir + Tipranavir
Time of maximum concentration (Tmax) | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
  14C-radiolabeled Tipranavir + Tipranavir
Apparent terminal half life (t1/2) | -10 minutes, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, and 12 hours after dose administration
  14C-radiolabeled Tipranavir + Tipranavir
Cumulative amount of 14C- radioactivity in Urine and feces | up to 15 days
Percent excretion in urine and feces | up to 15 days
  relative to total radioactivity administered
Time needed to achieve steady-state as determined by tipranavir trough concentrations | up to 15 days

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 15 days
Number of subjects with abnormal changes in laboratory parameters | up to day 14
Number of subjects with clinically significant changes in Electrocardiogram (ECG) | up to day 6